CLINICAL TRIAL: NCT03729388
Title: Treatment for Opiate Addiction: Prognostic fActors of Responsiveness to Maintenance Treatment
Acronym: TOPAZE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: CSAPA Apsyades (Unknown); OPPELIA-Le triangle (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC17_0377
Record Dates: First submitted 2018-10-04; First posted 2018-11-02 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Opioid-use Disorder
Keywords: Opiate substitution treatment; Opioid-related disorder; Behavior; Addictive; Substance-related disorder; Methadone; Buprenorphine; Prognosis
MeSH Terms: conditions — Opioid-Related Disorders; Behavior; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prognosis factor associated with good outcome. — Implementation of a systematic assessment of patient with OMT initiation. Patients included in the TOPAZE study will receive standardized clinical interviews, electrocardiograms, urinary and blood tests during a 12 months follow-up.

SUMMARY:
A global and integrative treatment of opioid-use disorders (OUD) with opiate maintenance therapy (OMT) and psychosocial interventions is recommended by all current guidelines. Treatment of OUD aim at prevents risks and consequences of opioid use (death by overdose, contamination with infectious diseases, mental and physical degradation, social exclusion and decrease of quality of life). OMT are approved since more than 20 years for OUD and a large number of patients have been treated. Nevertheless, identification of prognosis factors associated with good outcome is still limited. OMT duration, high dosages of OMT and patient good consistency have been identified as good prognosis factors but other individual factors could be involved and explain why OMT isn't as effective for all patients. The investigators assume that social environment, other addictive behaviors, psychiatric comorbidities, personality disorders and pharmacogenetics parameters might be of interest. Association between phenotype/ genotype, safety of OMT and therapeutic outcome will be especially assessed. For voluntary patients specific tools for risk reduction will be implemented (screening of infectious diseases with blood tests and fibrosis with fibroscan). Thus, the aim of TOPAZE study is to highlight prognosis factors for good outcome in the treatment of OUD moderate to severe at 12 months follow-up. Three main axes will be considered: clinical, pharmacological and pharmacogenetics.

DETAILED DESCRIPTION:
All patients with moderate or severe OUD diagnosis (according to Diagnostic and Statistical Manual Diploma in Social Medicine 5) who initiate OMT in addictionology department of Nantes hospital or in addiction care and prevention centers of Nantes could be included. Data will be collected during 3 visits.

During the first visit (inclusion), clinical interview, electrocardiogram, urinary and blood tests (pharmacokinetics and pharmacogenetics analysis) will be provided. Infectious disease screening and fibroscan could be also provided as the patient wishes. Inclusion visit will also correspond to initiation of OMT.

At 6 months follow-up (second visit) clinical interview, electrocardiogram, urinary and blood tests (pharmacokinetics and pharmacogenetics analysis) will be provided.

At 12 months follow-up (final visit) clinical interview, electrocardiogram and urinary test will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Initiation of treatment with OMT (methadone or buprenorphine) for an OUD moderate to severe (according to DSM 5) in Nantes Hospital addictionology department or in an addiction care and prevention centers in Nantes.
* Affiliated to social security
* Consent to participate

Exclusion Criteria:

* Upper cerebral function disorder inconsistent with participating in the study
* Difficulty to understand, read or write French language
* Adult under guardianship or curatorr
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include subjects with an opioid-related disorder for whom an OMT is indicated.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Clinical, pharmacokinetics and pharmacogenetics characteristics associated with good outcome of patients treated with OMT. | 12 months
  Good outcome is defined as early remission of opioid-related disorder according to Diagnostic and Statistical Manual of Mental Disorders Fifth version (none of the diagnostic criteria except craving within last three months) and no initiation or worsening of other addictive behavior (substance use disorders or gambling disorder according to Diagnostic and Statistical Manual of Mental Disorders Fifth version within last 12 months).

SECONDARY OUTCOMES:
Prevalence of good outcome after an OMT treatment initiation. | 12 months
  Good outcome is defined as early remission of opioid-related disorder according to Diagnostic and Statistical Manual of Mental Disorders Fifth version (none of the diagnostic criteria except craving within last three months) and no initiation or worsening of other addictive behavior (substance use disorders or gambling according to Diagnostic and Statistical Manual of Mental Disorders Fifth version within last 12 months).
Reasons for dropping-out of treatment. | 12 months
  Prevalence of each reason will be described (stopping treatment, death…).
Clinical characteristics of patients: history of psychoactive substance consumptions, psychiatric comorbidities and addictive behaviors, risky behaviors (intravenous administration, sharing equipment and sexual behavior). | 12 months
Number of participants with variation in the cytochrome P450 (CYP) enzyme with focus on CYP2B6, CYP2C19, CYP2D6, CYP3A4 polymorphisms using next-generation sequencing. | At inclusion
  Prevalence of CYP2B6, CYP2C19, CYP2D6 and CYP3A4 variants.
Pharmacokinetics of OMT elimination. | 6 months
  Residual plasmatic concentration will be considered.
Number of participants with methadone-associated Q-T interval prolongation as assessed by electrocardiogram [safety]. | 12 months
  Prevalence of methadone-associated Q-T interval prolongation.
Number of participants who accept to participate to a specific consultation with a hepatologist with a formation in risk reduction. | At inclusion
  Prevalence of participants who accept the hepatologist consultation and to be tested with blood tests for viral infections and fibroscan for hepatic fibrosis.
Number of participants with variation of the Permeability-glycoProtein (P-gP) using next-generation sequencing. | At inclusion
  Prevalence of P-gP variants.
Number of participants with variation in the OPRM1 gene (coding for µ receptor) using next-generation sequencing. | At inclusion
  Prevalence of OPRM1 variants.
Number of participants with urine tests results in accordance with a good compliance [compliance]. | At inclusion
  Prevalence of participants with positive urine tests results for OMT without any positive urine tests results for illicit substances or drugs without prescription.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Grall Bronnec, Nantes
  - OPPELIA-Le triangle, Nantes

IPD SHARING:
Plan to Share IPD: Undecided